CLINICAL TRIAL: NCT06726655
Title: Patterns of Neonatal Seizures At Assiut University Children's Hospital
Brief Title: Patterns of Neonatal Seizures
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mamoud Sabra Ahmed Hafez, 71515,Assiut, Assiut University
Other Study IDs: Neonatal seizures
Record Dates: First submitted 2024-12-06; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-10

CONDITIONS: Neonatal Seizures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Study the pattern of neonatal seizures in neonatal intensive care unit at Assiut university children's hospital along year from (Oct.2025-Oct.2026)

DETAILED DESCRIPTION:
Neonatal seizures are a commonly encountered neurologic condition in neonates.[1][2][3] They are defined as the occurrence of sudden, paroxysmal, abnormal alteration of electrographic activity at any point from birth to the end of the neonatal period[3]. This can be due to excessive excitatory or deficient inhibitory neuronal discharges.[1][4] Due to its immature state, the neonatal brain is prone to seizures due to an imbalance of neuronal excitation over inhibition.[1] The incidence has been reported between 1 to 5.5 per 1000 live births in term infants, with higher incidences reported in preterm infants[5]][6][7].

The classification of neonatal seizure as follows

Subtle Seizures:

They imitate normal behaviours and reactions like the following Ocular movements and Oral-buccal-lingual movements

Motor Seizures:

Clonic seizures are rhythmic jerks that may localise in a small part of the face or limbs, axial muscles and the diaphragm or be multifocal or hemiconvulsive.

Tonic seizures manifest with sustained contraction of facial, limb, axial and other muscles. They may be focal, multifocal or generalised, symmetrical or asymmetrical. Truncal or limb tonic extension imitates decerebrate or decorticate posturing.

Myoclonic seizures are rapid, single or arrhythmic repetitive jerks. They may affect a finger, a limb or the whole body. They may mimic the Moro reflex and startling responses.

Spasms producing flexion or extension similar to those of West syndrome are rare.

Autonomic Ictal Manifestations:

These are paroxysmal changes of heart rate, respiration, systemic blood pressure and apnea[8][9] Management include management of the cause and therapeutic hypothermia for hypoxic-ischemic encephalopathy[10], antibiotics for sepsis/meningitis, providing dextrose if the patient is severely hypoglycemic, correction of electrolyte abnormalities, or referral to neurosurgery if the patient has evidence of an intracranial hemorrhage. If the patient is suspected of having an inborn error of metabolism, halting of feeds, correcting metabolic derangements, and empiric therapy with vitamin and cofactor replacement may be initiated.[6][11][12] If the seizure is clinically evident and prolonged, the most common first-line agent utilized is phenobarbital.[13][14] If seizures do not resolve after the first loading dose, repeat boluses of this medication should be given. The next agent commonly utilized is fosphenytoin.[15] Other agents include levetiracetam and lidocaine in selected settings.[14] Short-acting benzodiazepines (i.e., midazolam) can be utilized if there is a delay in administering these agents.

The prognosis of neonatal seizures depends on the underlying etiology. If EEG is normal the prognosis is excellent but if EEG has many abnormalities such neonates have a poor prognosis and may develop cerebral palsy and epilepsy.The mortality rate of neonatal seizures is reported to be as high as 20%.[13] In survivors, neurologic impairment, disability, developmental delay, and epilepsy are common.[16][17][18][19]

ELIGIBILITY:
Inclusion criteria:

Study population comprised of term and preterm newborns who suffered from neonatal seizures.

Exclusion Criteria:

* Neoborns presented with non-epileptic behaviors include sucking movements, hiccuping, and benign neonatal sleep myoclonus (physiologic myoclonus that occurs during sleep). Motor automatisms (i.e., repetitive eye-opening, eye deviation, repetitive mouth, and tongue movements, bicycling of the lower extremities, tonic posturing).

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: all neonates comes to Assiut University Hospital with convulsions
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Study the pattern of neonatal seizures in neonatal intensive care unit at Assiut university children's hospital along year from (Oct.2025-Oct.2026) | along one year from (Oct.2025-Oct.2026)

REFERENCES:
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3925308/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/23622196/